CLINICAL TRIAL: NCT05269303
Title: Optimizing the Health-related Functions of a Wearable Monitoring Device in the Daily Life of Community-dwelling Older Adults: A Randomized Pilot Study
Brief Title: Wearable Monitoring Device in Daily Lives of Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Assistant professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A001523
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Device Ineffective
Keywords: community-dwelling older adults; Wearable monitoring device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive a 3-month Live With Wearable Monitoring Device program.
  Interventions: Device: Live With Wearable Monitoring Device program
- Control group (No Intervention): Usual care. As with the participants in the intervention group, those in the control group can utilize the features in the Wearable Monitoring Device.

INTERVENTIONS:
Device: Live With Wearable Monitoring Device program — The participants in the intervention group will receive a home visit by a Community Healthcare Worker in the first month, and biweekly motivational messages via Whats App in the second and third months.
  Arms: Intervention group

SUMMARY:
The aim is to implement an intervention program to promote the continued use of Wearable Monitoring Devices among older adults through a peer support approach facilitating the incorporation of Wearable Monitoring Devices in daily life.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* own a smartphone
* able to communicate in Cantonese or Mandarin
* able to access the Internet at home or elsewhere

Exclusion Criteria:

* have a confirmed diagnosis of cognitive impairment
* bed-bound
* currently own a wearable monitoring device
* have already engaged in other wearable device studies

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
The change of use intention of wearable monitoring device | Data collection will be conducted at the 1-month (T1), 3-month (T2), and 6-month (T3) time points
  It will be measured using a 4-item, 5-point Likert scale adopted from Bhattacherjee (2001) and Windasari et al. (2021). The five-point scale ranges from 1 = not at all satisfied to 5 = very certain, with higher scores representing a higher chance of continuing to use the WMD.

SECONDARY OUTCOMES:
The change of adherence rate of wearing wearable monitoring device | Data collection will be conducted at the 1-month (T1), 3-month (T2), and 6-month (T3) time points
  It will be measured by checking in our database the number of days that participants wore their device, and the average amount of time worn per day. Longer time worn represents better adherence rate
The change in quality of life among baseline (T0) and at the 1-month (T1), 3-month (T2), and 6-month (T3) time points | baseline (T0) and at the 1-month (T1), 3-month (T2), and 6-month (T3) time points
  Quality of life will be measured using the Hong Kong version of the EuroQol 5-dimension scale. The EQ-5D-5L is comprised of five dimensions, namely, mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. The utility score ranges from 0 to 1, with higher means better quality of life
The change of health service utilization among baseline (T0) and at the 1-month (T1), 3-month (T2), and 6-month (T3) time points | baseline (T0) and at the 1-month (T1), 3-month (T2), and 6-month (T3) time points
  ealth service utilization includes the number of attendances at a general practitioner's office, emergency department, hospital, and general out-patient clinic. The data will be reported by the participants and confirmed with medical and attendance certificates
Recruitment rate | baseline pre-intervention
  The recruitment rate will be calculated by dividing the number of participants who are recruited and randomized, by the number of eligible participants.
Attrition rate | 6-month (T3) time points
  The attrition rate refers to the number of participants who withdraw from the study or who are lost to follow up.
Incidence of reports of adverse events | 6-month (T3) time points
  the incidence of reports of adverse events will be recorded by a staff member assigned to each of the community centres and a nurse
Incidence of reports of technical difficulties | 6-month (T3) time points
  Incidence of reports of technical difficulties will be recorded by a staff member assigned to each of the community centres and a nurse
The change of perceived usability of the wearable monitoring device before and after the program | baseline pre-intervention, 6-month (T3) time points
  The participants will be required to complete a questionnaire that measures their attitude towards using the WMD; the perceived usefulness, perceived ease of use, and self-efficacy of using the device; and their level of anxiety about using the device. The questionnaire was drawn up by Chen and Chan (2014). This 10-point Likert scale ranges from 1 (strongly disagree) to 10 (strongly agree), with higher marks indicating a better outcome, with the exception of the item on anxiety levels, where higher marks represent a higher level of anxiety in using the WMD.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, Ph.D., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Siu Sai Wan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AKC, Bayuo J, Su JJ, Wong FKY, Chow KKS, Wong BP, Wong SM, Hui V. Effectiveness of the Support From Community Health Workers and Health Care Professionals on the Sustained Use of Wearable Monitoring Devices Among Community-Dwelling Older Adults: Feasibility Randomized Controlled Trial. J Med Internet Res. 2024 Nov 18;26:e52435. doi: 10.2196/52435. PMID 39556810
- [Derived] Wong AKC, Tso WC, Su JJ, Hui VCC, Chow KKS, Wong SM, Wong BB, Wong FKY. Effectiveness of support from community health workers on the sustained use of a wearable monitoring device among community-dwelling older adults: A randomized trial protocol. PLoS One. 2023 Dec 22;18(12):e0294517. doi: 10.1371/journal.pone.0294517. eCollection 2023. PMID 38134126